CLINICAL TRIAL: NCT06831344
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 5-Period Crossover Study to Determine the Bioavailability of Two Vonoprazan Orally Disintegrating Tablet Formulations Administered Without Water or Mixed With Water and Administered Via a Syringe Relative to the Vonoprazan Tablet in Healthy Subjects
Brief Title: A Study to Evaluate Two Vonoprazan Orally Disintegrating Tablet Formulations Administered Without Water or Mixed With Water and Administered Via a Syringe Relative to the Vonoprazan Tablet in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VPED-105
Record Dates: First submitted 2025-02-14; First posted 2025-02-18 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Erosive Esophagitis; Non-erosive Gastroesophageal Reflux Disease; Vonoprazan
MeSH Terms: interventions — Water; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Intervention Model Description: The treatment periods will include administration of single doses of vonoprazan 10 mg on Day 1 of each period. There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sequence A, B, C, D, E: Vonoprazan 10 mg (Experimental): Participants will be randomly assigned to 1 of 5 treatment sequences in a 1:1:1:1:1 ratio.
  On the first day of each dosing period, participants will receive 1 of the following study treatments according to the treatment sequence they are randomly assigned to:
  * Treatment A: Vonoprazan 10 mg ODT-1 without water
  * Treatment B: Vonoprazan 10 mg ODT-1 mixed with water and administered via a syringe
  * Treatment C: Vonoprazan 10 mg ODT-2 without water
  * Treatment D: Vonoprazan 10 mg ODT-2 mixed with water and administered via a syringe
  * Treatment E (reference): Vonoprazan 10 mg tablet.
  There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
  Interventions: Drug: Vonoprazan ODT-1 or ODT-2 without Water; Drug: Vonoprazan ODT-1 or ODT-2 with Water; Drug: Vonoprazan (Reference)
- Sequence B, D, E, C, A: Vonoprazan 10 mg (Experimental): Participants will be randomly assigned to 1 of 5 treatment sequences in a 1:1:1:1:1 ratio.
  On the first day of each dosing period, participants will receive 1 of the following study treatments according to the treatment sequence they are randomly assigned to:
  * Treatment A: Vonoprazan 10 mg ODT-1 without water
  * Treatment B: Vonoprazan 10 mg ODT-1 mixed with water and administered via a syringe
  * Treatment C: Vonoprazan 10 mg ODT-2 without water
  * Treatment D: Vonoprazan 10 mg ODT-2 mixed with water and administered via a syringe
  * Treatment E (reference): Vonoprazan 10 mg tablet.
  There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
  Interventions: Drug: Vonoprazan ODT-1 or ODT-2 without Water; Drug: Vonoprazan ODT-1 or ODT-2 with Water; Drug: Vonoprazan (Reference)
- Sequence C, E, B, A, D: Vonoprazan 10 mg (Experimental): Participants will be randomly assigned to 1 of 5 treatment sequences in a 1:1:1:1:1 ratio.
  On the first day of each dosing period, participants will receive 1 of the following study treatments according to the treatment sequence they are randomly assigned to:
  * Treatment A: Vonoprazan 10 mg ODT-1 without water
  * Treatment B: Vonoprazan 10 mg ODT-1 mixed with water and administered via a syringe
  * Treatment C: Vonoprazan 10 mg ODT-2 without water
  * Treatment D: Vonoprazan 10 mg ODT-2 mixed with water and administered via a syringe
  * Treatment E (reference): Vonoprazan 10 mg tablet.
  There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
  Interventions: Drug: Vonoprazan ODT-1 or ODT-2 without Water; Drug: Vonoprazan ODT-1 or ODT-2 with Water; Drug: Vonoprazan (Reference)
- Sequence D, C, A, E, B: Vonoprazan 10 mg (Experimental): Participants will be randomly assigned to 1 of 5 treatment sequences in a 1:1:1:1:1 ratio.
  On the first day of each dosing period, participants will receive 1 of the following study treatments according to the treatment sequence they are randomly assigned to:
  * Treatment A: Vonoprazan 10 mg ODT-1 without water
  * Treatment B: Vonoprazan 10 mg ODT-1 mixed with water and administered via a syringe
  * Treatment C: Vonoprazan 10 mg ODT-2 without water
  * Treatment D: Vonoprazan 10 mg ODT-2 mixed with water and administered via a syringe
  * Treatment E (reference): Vonoprazan 10 mg tablet.
  There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
  Interventions: Drug: Vonoprazan ODT-1 or ODT-2 without Water; Drug: Vonoprazan ODT-1 or ODT-2 with Water; Drug: Vonoprazan (Reference)
- Sequence E, A, D, B, C: Vonoprazan 10 mg (Experimental): Participants will be randomly assigned to 1 of 5 treatment sequences in a 1:1:1:1:1 ratio.
  On the first day of each dosing period, participants will receive 1 of the following study treatments according to the treatment sequence they are randomly assigned to:
  * Treatment A: Vonoprazan 10 mg ODT-1 without water
  * Treatment B: Vonoprazan 10 mg ODT-1 mixed with water and administered via a syringe
  * Treatment C: Vonoprazan 10 mg ODT-2 without water
  * Treatment D: Vonoprazan 10 mg ODT-2 mixed with water and administered via a syringe
  * Treatment E (reference): Vonoprazan 10 mg tablet.
  There will be a washout interval of a minimum of 5 days between study drug dosing in each period.
  Interventions: Drug: Vonoprazan ODT-1 or ODT-2 without Water; Drug: Vonoprazan ODT-1 or ODT-2 with Water; Drug: Vonoprazan (Reference)

INTERVENTIONS:
Drug: Vonoprazan ODT-1 or ODT-2 without Water — Vonoprazan will be administered orally as an ODT-1 or ODT-2 without water
Drug: Vonoprazan ODT-1 or ODT-2 with Water — Vonoprazan will be administered orally as an ODT-1 or ODT-2 with water via a syringe
Drug: Vonoprazan (Reference) — Vonoprazan will be administered orally as a tablet

SUMMARY:
The primary objective of this study is to assess the bioavailability (BA) of a single oral dose of two vonoprazan orally disintegrating tablet formulations (ODT-1 or ODT-2) administered without water or mixed with water and administered via a syringe relative to the vonoprazan tablet in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 18 to 55 years of age, inclusive, at Screening.
* The participant has a body mass index (BMI) 18 to 32 kg/m2, inclusive, at Screening.
* The participant is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at Screening.
* Female participants of reproductive potential must use an acceptable method of birth control (ie, diaphragm with spermicide, intrauterine device, condom with foam or vaginal spermicide, oral contraceptives, or abstinence) from signing the informed consent form (ICF) until 4 weeks after the last dose of study drug or be surgically sterile (ie, hysterectomy or bilateral oophorectomy) or postmenopausal (defined as amenorrhea for 12 consecutive months and documented plasma follicle stimulating hormone [FSH] level >40 IU/mL during Screening).
* Female participants must have a negative pregnancy test at Screening and upon Check-in.
* The participant agrees to comply with all protocol requirements.
* The participant is able to provide written informed consent.

Exclusion Criteria:

* The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies at Screening.
* The participant has a positive test result for the presence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Check-in.
* The participant has a history of a clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality that may impact the ability of the subject to participate.
* The participant has current or recent (within 6 months) gastrointestinal conditions that would be expected to influence the absorption of drugs (eg, history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis (EE)), frequent (more than once per week) occurrence of heartburn, or any surgical intervention.
* The participant has any other clinically significant findings on physical examination, clinical laboratory abnormalities, and/or ECG results that preclude his/her participation in the study, as deemed by the investigator.
* The participant has used any prescription (excluding hormonal birth control) and/or over-the-counter medications (including Cytochrome P450 3A4 (CYP3A4) inducers) except acetaminophen (up to 2 g per day), including herbal or nutritional supplements, within 14 days before the first dose of study drug, and/or is expected to require any such medication during the course of the study until the end of confinement on Study Day 23.
* The participant has consumed grapefruit and/or grapefruit juice, Seville orange or Seville orange-containing products (eg, marmalade), or other food products that may be CYP3A4 inhibitors (eg, vegetables from the mustard green family [kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 7 days before the first dose of study drug and/or is expected to be unable to abstain through the study.
* The participant has consumed caffeine- or xanthine-containing products within 48 hours (or 5 half-lives) before the first dose of study drug and/or is unable to abstain through the study.
* The participant is a smoker and/or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* The participant has a history of alcohol abuse and/or drug addiction within the last year or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects; 1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits) or use of alcohol 48 hours before the first dose of study drug.
* The participant has a positive test result for drugs of abuse, alcohol, or cotinine (indicating active current smoking) at Screening or Check-in.
* The participant is involved in strenuous activity or contact sports within 24 hours before the first dose of study drug and during the study.
* The participant has donated blood or blood products >450 mL within 30 days before the first dose of study drug.
* The participant has a history of relevant drug and/or food allergies (ie, allergy to vonoprazan or excipients or any significant food allergy that could preclude a standard diet in the clinical unit).
* The participant has received a study drug in another investigational study within 5-times the t1/2 of the study drug or 30 days of dosing, whichever is longer.
* Female participants who are pregnant or lactating; intend to become pregnant before, during, or within 4 weeks after participating in this study; or intend to donate ova during this time period.
* The participant is not suitable for entry into the study in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-04-05 (Actual); Study Completion 2025-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (1):
- 7551 Metro Center Dr Ste 200, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in the United States from 14 February 2025 to 10 April 2025.
Pre-assignment Details: A total of 25 healthy participants were enrolled in this 5-period crossover study and were randomized to 1 of 5 treatment sequences to receive vonoprazan as two formulations (orally dispersible tablet [ODT]-1 and ODT-2) with or without water. The reference formulation was vonoprazan 10 milligram (mg) tablets (Treatment E).
Groups:
- Vonoprazan 10 mg: Treatment Sequence 1: Participants received Vonoprazan 10 mg, orally, in the following sequence: ODT-1, once on Day 1 of Period 1 without water as Treatment A, ODT-1, once on Day 1 of Period 2 mixed with water and administered via a syringe as Treatment B, ODT-2, once on Day 1 of Period 3 without water as Treatment C, ODT-2, once on Day 1 of Period 4 mixed with water and administered via a syringe as Treatment D, and Vonoprazan 10 mg tablet, once on Day 1 of Period 5 as Treatment E. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between doses in each treatment period.
- Vonoprazan 10 mg: Treatment Sequence 2: Participants received Vonoprazan 10 mg, orally, in the following sequence: ODT-1, once on Day 1 of Period 1 mixed with water and administered via a syringe as Treatment B, ODT-2, once on Day 1 of Period 2 mixed with water and administered via a syringe as Treatment D, Vonoprazan 10 mg tablet, once on Day 1 of Period 3 as Treatment E, ODT-2, once on Day 1 of Period 4 without water as Treatment C, ODT-1, and once on Day 1 of Period 5 without water as Treatment A. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between doses in each treatment period.
- Vonoprazan 10 mg: Treatment Sequence 3: Participants received Vonoprazan 10 mg, orally, in the following sequence: ODT-2, once on Day 1 of Period 1 without water as Treatment C, Vonoprazan 10 mg tablet, once on Day 1 of Period 2 as Treatment E, ODT-1, once on Day 1 of Period 3 mixed with water and administered via a syringe as Treatment B, ODT-1, once on Day 1 of Period 4 without water as Treatment A and ODT-2, once on Day 1 of Period 5 mixed with water and administered via a syringe as Treatment D. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between doses in each treatment period.
- Vonoprazan 10 mg: Treatment Sequence 4: Participants received Vonoprazan 10 mg, orally, in the following sequence: ODT-2, once on Day 1 of Period 1 mixed with water and administered via a syringe as Treatment D, ODT-2, once on Day 1 of Period 2 without water as Treatment C, ODT-1, once on Day 1 of Period 3 without water as Treatment A, Vonoprazan 10 mg tablet, once on Day 1 of Period 4 as Treatment E and ODT-1, once on Day 1 of Period 5 mixed with water and administered via a syringe as Treatment B. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between doses in each treatment period.
- Vonoprazan 10 mg: Treatment Sequence 5: Participants received Vonoprazan 10 mg, orally, in the following sequence: Vonoprazan 10 mg tablet, once on Day 1 of Period 1 as Treatment E, ODT-1, once on Day 1 of Period 2 without water as Treatment A, ODT-2, once on Day 1 of Period 3 mixed with water and administered via a syringe as Treatment D, ODT-1, once on Day 1 of Period 4 mixed with water and administered via a syringe as Treatment B and ODT-2, once on Day 1 of Period 5 without water as Treatment C. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between doses in each treatment period.
Period: Overall Study
Arm/Group | Vonoprazan 10 mg: Treatment Sequence 1 | Vonoprazan 10 mg: Treatment Sequence 2 | Vonoprazan 10 mg: Treatment Sequence 3 | Vonoprazan 10 mg: Treatment Sequence 4 | Vonoprazan 10 mg: Treatment Sequence 5
Started | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who receive at least 1 dose of study drug. As planned, baseline data was collected and reported as single arm for all 25 participants.
Groups:
- All Participants: All participants who were randomized to receive Vonoprazan 10 mg, orally, in one of the five treatment sequence: ODT-1, once on Day 1 of Period 1 without water as Treatment A, ODT-1, once on Day 1 of Period 2 mixed with water and administered via a syringe as Treatment B, ODT-2, once on Day 1 of Period 3 without water as Treatment C, ODT-2, once on Day 1 of Period 4 mixed with water and administered via a syringe as Treatment D, and Vonoprazan 10 mg tablet, once on Day 1 of Period 5 as Treatment E. Each treatment period was 3 days, with treatment received on Day 1 of each treatment period. A washout interval of minimum of 5 days was maintained between each treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Drug Concentration (Cmax) of Vonoprazan
Description: Cmax of Vonoprazan was reported.
Time Frame: Day 1 of each 3-day treatment period: Within 15 minutes pre-dose and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours post-dose
Population: The Pharmacokinetic (PK) population included participants who received at least 1 dose of study drug and had sufficient concentration data to support accurate estimation of at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: Vonoprazan 10 mg: Participants received Vonoprazan 10 mg ODT-1 tablets, orally, once on Day 1 of the allocated period without water.
- Treatment B: Vonoprazan 10 mg: Participants received Vonoprazan 10 mg ODT-1 tablets, orally, once on Day 1 of the allocated period mixed with water and administered via a syringe.
- Treatment C: Vonoprazan 10 mg: Participants received Vonoprazan 10 mg ODT-2 tablets, orally, once on Day 1 of the allocated period without water.
- Treatment D: Vonoprazan 10 mg: Participants received Vonoprazan 10 mg ODT-2 tablets, once on Day 1 of the allocated period mixed with water and administered via a syringe.
- Treatment E: Vonoprazan 10 mg: Participants received Vonoprazan 10 mg tablets, orally, once on Day 1 of the allocated period.
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
nanogram per milliliter (ng/mL) | 6.11 (47.8) | 5.81 (41.4) | 5.46 (36.1) | 5.72 (46.2) | 5.40 (38.4)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — The two treatments were deemed equivalent if the 90% confidence intervals (CIs) for the geometric mean ratios (GMRs) for all of the parameters were each within 80.00% and 125.00%; Ratio of GLSM Percentage (%) = 113.26, 90% CI 2-sided [104.86 to 122.33] — Geometric least square mean (GLSM) ratios were calculated by taking antilog of difference of least square means and associated 90% confidence intervals (CIs) from linear mixed effect model analyzing natural logarithms of corresponding PK parameters
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — The two treatments were deemed equivalent if the 90% CIs for the GMRs for all of the parameters were each within 80.00% and 125.00%; Ratio of GLSM (%) = 107.65, 90% CI 2-sided [99.67 to 116.28] — GLSM ratios were calculated by taking the antilog of the difference of least square means and associated 90% CIs from the linear mixed effect model analyzing the natural logarithms of the corresponding PK parameters
Statistical Analysis 3: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 101.19, 90% CI 2-sided [93.68 to 109.30] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Treatment D: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 105.94, 90% CI 2-sided [98.08 to 114.43] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment B: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 95.05, 90% CI 2-sided [88.00 to 102.67] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment D: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 104.69, 90% CI 2-sided [96.93 to 113.08] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-t) of Vonoprazan
Description: AUC0-t of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: The PK population included participants who received at least 1 dose of study drug and had sufficient concentration data to support accurate estimation of at least 1 PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*hour/mL | 57.1 (45.8) | 54.8 (42.0) | 52.8 (41.7) | 51.7 (47.6) | 49.8 (38.5)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 114.62, 90% CI 2-sided [107.46 to 122.24] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 110.01, 90% CI 2-sided [103.14 to 117.33] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 106.00, 90% CI 2-sided [99.39 to 113.06] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Treatment D: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 103.87, 90% CI 2-sided [97.39 to 110.78] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment B: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 95.98, 90% CI 2-sided [89.99 to 102.37] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment D: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 97.99, 90% CI 2-sided [91.87 to 104.51] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: AUC From Time 0 Extrapolated to Infinity (AUC0-inf) of Vonoprazan
Description: AUC0-inf of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
ng*hour/mL | 59.2 (44.3) | 57.1 (39.4) | 55.3 (39.0) | 54.1 (44.9) | 51.9 (36.3)
Statistical Analysis 1: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 114.01, 90% CI 2-sided [107.28 to 121.17] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Treatment B: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 109.99, 90% CI 2-sided [103.49 to 116.90] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 106.55, 90% CI 2-sided [100.26 to 113.24] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Treatment D: Vonoprazan 10 mg vs Treatment E: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 104.31, 90% CI 2-sided [98.15 to 110.86] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Treatment A: Vonoprazan 10 mg vs Treatment B: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 96.47, 90% CI 2-sided [90.77 to 102.53] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Treatment C: Vonoprazan 10 mg vs Treatment D: Vonoprazan 10 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; Ratio of GLSM (%) = 97.90, 90% CI 2-sided [92.11 to 104.05] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Vonoprazan
Description: Tmax of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hours | 2.00 [1.50 to 6.00] | 2.00 [1.50 to 6.00] | 2.12 [1.50 to 4.08] | 2.00 [1.50 to 6.00] | 2.00 [1.00 to 6.00]

5. Secondary Outcome: Time Until First Measurable Concentration in Plasma (Tlag) of Vonoprazan
Description: Tlag of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hours | 0.32 [0.25 to 1.02] | 0.25 [0.25 to 1.00] | 0.32 [0.25 to 1.00] | 0.25 [0.25 to 1.50] | 0.27 [0.25 to 1.50]

6. Secondary Outcome: Terminal Elimination Rate Constant (λz) of Vonoprazan
Description: λz of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
per hour | 0.0948 (0.0175) | 0.0998 (0.0188) | 0.0955 (0.0167) | 0.0963 (0.0140) | 0.0975 (0.0185)

7. Secondary Outcome: Terminal Phase Half-life (t1/2) of Vonoprazan
Description: t1/2 of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
hours | 7.54 (1.36) | 7.20 (1.42) | 7.48 (1.38) | 7.36 (1.22) | 7.35 (1.36)

8. Secondary Outcome: Apparent Oral Clearance (CL/F) of Vonoprazan
Description: CL/F of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: litres/hour (L/h)
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
litres/hour (L/h) | 184 (78.9) | 188 (76.0) | 193 (72.5) | 202 (89.2) | 205 (75.9)

9. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Vonoprazan
Description: Vz/F of Vonoprazan was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: litres (L)
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
litres (L) | 1930 (735) | 1880 (622) | 2030 (678) | 2070 (762) | 2100 (668)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 28
Description: All-cause mortality, serious and non-serious adverse events were measured in the safety population, which included all participants who received at least 1 dose of study drug. Safety data are presented for each treatment received, as pre-specified.
Arm/Group | Treatment A: Vonoprazan 10 mg | Treatment B: Vonoprazan 10 mg | Treatment C: Vonoprazan 10 mg | Treatment D: Vonoprazan 10 mg | Treatment E: Vonoprazan 10 mg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 0/25 | 1/25 | 1/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Vonoprazan 10 mg (N=25) | Treatment B: Vonoprazan 10 mg (N=25) | Treatment C: Vonoprazan 10 mg (N=25) | Treatment D: Vonoprazan 10 mg (N=25) | Treatment E: Vonoprazan 10 mg (N=25)
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) are not permitted to publish the data. Data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the PIs to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority over all such issues.

DOCUMENTS (2):
  • Study Protocol (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT06831344/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT06831344/SAP_001.pdf